CLINICAL TRIAL: NCT02915822
Title: COSMIC Study - Comparing Open Scarf/Akin Osteotomy and Minimally Invasive Chevron/Akin. A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181137
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimally Invasive Chevron/Akin osteotomy (Experimental): Minimally invasive technique to surgically correct Hallux Valgus
  Interventions: Procedure: Minimally Invasive Chevron/Akin osteotomy
- Open Scarf/Akin osteotomy (Active Comparator): Open technique to surgically correct Hallux Valgus
  Interventions: Procedure: Open Scarf/Akin osteotomy

INTERVENTIONS:
Procedure: Minimally Invasive Chevron/Akin osteotomy — Minimally invasive technique for hallux valgus correction
  Arms: Minimally Invasive Chevron/Akin osteotomy
Procedure: Open Scarf/Akin osteotomy — Open technique for Hallux Valgus correction
  Arms: Open Scarf/Akin osteotomy

SUMMARY:
The aim of this study is to assess the feasibility of conducting a study to compare the patient recorded and clinical outcomes for the surgical management of Hallux Valgus correction. A prospective trial will randomise the patients into two groups - Open Scarf/Akin osteotomy and Minimally Invasive Chevron/Akin osteotomy.

DETAILED DESCRIPTION:
This study will assess the feasibility of a prospective trial that would randomise the patients into two groups for surgical correction of Hallux Valgus - Open Scarf/Akin osteotomy and Minimally Invasive Chevron/Akin osteotomy. Patients will complete a validated questionnaire (Manchester Oxford Foot questionnaire) preoperatively and post operatively at 6 months and 1 year. Range of motion of the Great Toe Metatarsal Phalangeal Joint will also be measured by goniometer. This study will assess the ability to recruit and retain patients and thus determine if a study comparing the surgical techniques would be feasible. In addition, for data collected statistical differences of the change in patient reported outcomes, range of motion between the two groups will be calculated with a significance level of p<0.05. This study will assess if a larger study comparing minimally invasive to open Hallux Valgus correction would be able to be performed

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with Hallux valgus deformity suitable for treatment by both Open Scarf/Akin and MICA procedures.
* Patients with no significant co-morbidities that would increase their risk of procedure.
* Patients able to understand and complete questionnaires.
* Patients with the capacity to provide informed consent.
* Patients who have, in addition to Hallux Valgus Deformity, lesser toe deformities requiring correction distal to the metatarsal phalangeal joint at time of procedure.
* Patients without significant other mid foot or hind foot pathology

Exclusion Criteria:

* Patients under 18 years of age
* Patients with severity of Hallux valgus deformity necessitating Open procedure
* Patients with significant co-morbidities that would increase the risk of surgery
* Patients unable to understand or complete questionnaires.
* Patients without the capacity to provide informed consent.
* Patients with additional deformity requiring additional procedures proximal to the metatarsal phalangeal joint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2023-03-05 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Number of patients recruited | 1 year
  The number of patients able to be recruited and retained in this feasibility study. This will determine if a larger study can go forward.

SECONDARY OUTCOMES:
Patient reported outcomes assessed by questionnaire | 1 year
  Patient satisfaction, MOXFQ score recorded by questionnaire preoperatively, at 6 months and at 1 year.
MTPJ range of movement in degrees | 6 months
  Measured preoperatively at 6 weeks and 6 months by goniometer
Complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rajeshkumar Kakwani, Study Chair — Northumbria Healthcare NHS Trust
Locations (1):
- Northumbria NHS Foundation Trust, Newcastle upon Tyne, Northumbria, United Kingdom

IPD SHARING:
Plan to Share IPD: No